CLINICAL TRIAL: NCT05695404
Title: Contribution of 3D Printing in Anatomical Lung Segmentectomies: a Prospective Randomized Controlled Pilot Trial.
Brief Title: Contribution of 3D Printing in Anatomical Lung Segmentectomies.
Acronym: 3DiLUNG
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Fondation de l'Avenir (Other); Paris cite university, 75006 Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: THOR-02-2019
Record Dates: First submitted 2023-01-02; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Thoracic Surgery
Keywords: Segmentectomy; Thoracic surgery; 3D printed model; Mental workload; 3D reconstruction
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The "Digital" arm: Surgeons had a virtual 3D reconstruction of the patient's pulmonary anatomy by the Visible Patient Planning (VP) software
  Interventions: Procedure: Segmentectomy
- The "Digital+Object" arm: Surgeons had at their disposal on the operating field, in a transparent sterile bag, the 3D printed model, made from the virtual 3D VP software of the patient's lung anatomy
  Interventions: Procedure: Segmentectomy

INTERVENTIONS:
Procedure: Segmentectomy — Lung resection

SUMMARY:
The aim of the present work was to evaluate if the presence on the operating field of a 3D printed personalized model of the pulmonary anatomy of a patient operated by full thoracoscopy for an anatomical segmentectomy, makes it possible to reduce the mental workload and the fatigue of the surgeon.

DETAILED DESCRIPTION:
Between 28.10.2020 and 05.10.2021, we successively included all anatomic segmentectomies performed by full thoracoscopy in our department, except for S6 segmentectomies, S4+5 left bisegmentectomy and patients for whom the time to surgery was considered too short to obtain the 3D printed model before surgery.

We performed a prospective randomized controlled pilot trial on 2 parallel arms:

* The "Digital" arm
* The "Digital+Object" arm.

ELIGIBILITY:
Inclusion Criteria:

* all anatomic segmentectomies performed by full thoracoscopy, except for S6 segmentectomies, S4+5 left bisegmentectomy and patients for whom the time to surgery was considered too short to obtain the 3D printed model before surgery.

Exclusion Criteria:

* S6 segmentectomies
* S4+5 left bisegmentectomy
* Patients for whom the time to surgery was considered too short to obtain the 3D printed model before surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all anatomic segmentectomies performed by full thoracoscopy in our department.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Surgeon's mental workload. | 1 day
  measure of mental workload by the NASA-TLX score at the end of the surgery: It is a multidimensional rating scale that has six bipolar dimensions: mental demand (MD); physical demand (PD); time demand (TD); self performance (P); effort (E); and frustration (F). The dimensions thus reflect tasks (DM, PD, TD), performance (P), and behavioral factors (E and F). NASA-TLX is calculated through a self-questionnaire, using 20-point visual analogue scales anchored by very low and very high. The test provides a global load score between zero and 100 and by sub-dimensions, higher scores indicating higher mental loads of subjective perceptions.

SECONDARY OUTCOMES:
The surgeon's stress during surgery | 1 day
  To assess stress, the surgeon wore a Holter device throughout the surgical procedure
Surgeon's attention to work by d2-R test | 1 day
  For the evaluation of the surgeon's attention to work at the end of the surgery, we used first d2-R test.
  Scoring of the d2-R test included the following: concentration performance (CC), which represents the capacity of concentration; total number of target items processed, included the omitted ones (CCT), which informs about the speed of processing the test; percentage of errors (E%) which is defined as (total number of errors x 100)/CCT, and reflects performance accuracy.
  These scores are standardized to standard score (NS), used by default for the computerized d2-R. The NS ranges from 20 to 80, with an average of 50. In the normal distribution scale of the d2-R test, 7% of the normative subjects scored under 35, 24% scored between 35 and 44, 38% scored between 45 and 55, 24% scored from 56 to 65 and 7% scored over 65. The scores are consider very weak, weak, mean, high and very high, respectively.
Surgeon's attention to work by EncephalApp Stroop test. | 1 day
  For the evaluation of the surgeon's attention to work at the end of the surgery, we used also EncephalApp Stroop test.
  The task has two components: "off" and "on" states. In the "off " state, the surgeon views a pound signs (###) presented in red, green, or blue, one at a time and has to respond as quickly as possible by touching the matching color of the stimulus to the colors displayed at the bottom of the screen. In the "on" state the subject has to accurately select the color of the word presented, which is actually the name of the color in discordant coloring. The specific outcomes of the EncephalApp Stroop test were: the total time for five correct runs in the "off " state (OffTime) and in the "on" state (OnTime); the number of runs needed to complete the five correct "off" runs and five correct "on" runs.
The surgeon's overall satisfaction at the end of the surgery. | 1 day
  To assess surgeon subjective satisfaction at the end of the surgery, we used a subjective satisfaction 5-point Likert scale
Duration of the surgical procedure | 1 day
  calculated from the skin incision to the completion of the segmentectomy

CONTACTS AND LOCATIONS:
Overall Officials: Madalina Grigoroiu, dr, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris (thoracic surgery department), Paris, France